CLINICAL TRIAL: NCT07338500
Title: Cardiovascular Effects of Music Versus Guided Mindfulness: A Randomized Crossover Study
Brief Title: Cardiovascular Effects of Music Versus Guided Mindfulness
Acronym: CMM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Kyle Greenway, Psychiatrist, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2026-4674
Record Dates: First submitted 2025-12-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Music Listening Intervention; Mindfulness-based Intervention
Keywords: Music; Mindfulness
MeSH Terms: interventions — Music Therapy; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention First (Experimental): Participants randomized to this arm will receive a 40-minute Music Listening intervention in the first period, followed by a 20-minute washout period, and then receive a 40-minute Guided Mindfulness intervention in the second period.
  Interventions: Other: Music; Other: Mindfulness
- Mindfulness Intervention First (Experimental): Participants randomized to this arm will receive a 40-minute Guided Mindfulness intervention in the first period, followed by a 20-minute washout period, and then receive a 40-minute Music Listening intervention in the second period.
  Interventions: Other: Music; Other: Mindfulness

INTERVENTIONS:
Other: Music — Participants will listen to a 40-minute playlist, curated by the research team, through noise-cancelling headphones. The playlist will simultaneously be played in the room through speakers.
Other: Mindfulness — Participants will engage in a structured mindfulness session led by a member of the research team with experience in mindfulness-based practices. To ensure consistency across sessions, a standardized script will be used, which incorporates body scan meditation, breath coherence, and a guided emotional awareness exercise.

SUMMARY:
The purpose of this study is to examine how listening to music compares to guided mindfulness in affecting blood pressure, heart rate, and feelings of anxiety in healthy adults. The investigators aim to determine whether one of these approaches is more effective in reducing these variables. Additionally, the study will explore whether personal traits or preferences, measured using questionnaires, influence how participants respond to music or mindfulness. Based on previous clinical findings, the researchers hypothesize that listening to music will lead to greater reductions in blood pressure and heart rate compared to guided mindfulness.

DETAILED DESCRIPTION:
Music and mindfulness-based practices, such as meditation and breathing exercises, are well-established non-pharmacological interventions known to positively influence both physiological and psychological health. They are utilized for their ability to reduce stress and promote relaxation by modulating autonomic nervous system activity, which in turn influences the cardiovascular system. This modulation has been associated with reductions in markers of physiological stress, such as blood pressure and heart rate.

Cardiovascular influences of music and mindfulness have been leveraged in numerous medical procedures for enhancing comfort and tolerability, as well as mental well-being. However, despite the widespread use and documented physiological effects of music and mindfulness-based interventions, there is a lack of research directly comparing their effects. Furthermore, there is a relative lack of high-quality randomized trials examining the effects of music and mindfulness on parameters such as blood pressure and heart rate.

This randomized crossover study will examine the cardiovascular impact of listening to a curated music playlist versus participating in a guided mindfulness session in a healthy population to determine whether music produces greater reductions in blood pressure and heart rate than guided mindfulness.

Each participant will attend a single 3-hour study visit, during which they will take part in two sessions. One session involves listening to a carefully selected music playlist, and the other involves participating in a guided mindfulness exercise. The order of the sessions will be random. Blood pressure and heart rate will be measured throughout the study visit, and participants will be asked to complete questionnaires measuring anxiety, experience with music and mindfulness, tendency to become deeply engaged, and enjoyment of each session.

The primary aim is to compare changes in systolic blood pressure, diastolic blood pressure, and heart rate between curated music playlist and guided mindfulness interventions, using an automated oscillometric upper arm blood pressure monitor with measurements taken at 5-minute intervals.

By investigating the physiological effects of music versus guided mindfulness on hemodynamic responses in a healthy population, this study will provide critical insight into the distinct and shared autonomic effects of these two non-pharmacological interventions. Understanding the cardiovascular effects of music and guided mindfulness will inform evidence-based guidelines for integrating these interventions into clinical and research protocols. As non-invasive therapeutic tools, both music and mindfulness hold promise for enhancing patient care across diverse settings.

ELIGIBILITY:
Inclusion Criteria:

* Normal baseline blood pressure (systolic BP < 120 mmHg and diastolic BP < 80mmHg).
* Abstention from caffeine intake for at least 12 hours before the study session and throughout the session, as caffeine may influence cardiovascular measurements.
* Abstention from using nicotine or tobacco products for at least 1 hour before the study session and throughout the session, as these substances may influence cardiovascular measurements.

Exclusion Criteria:

* Significant hearing impairments that cannot be improved with hearing aids or sound amplification.
* Current use of medications that could affect blood pressure.
* History of hypertension or cardiovascular disease.
* Diagnosis of active substance use disorder, or reported patterns of alcohol, cannabis, or recreational/non-prescribed substance use likely to affect cardiovascular function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Changes in Blood Pressure | 0, 5, 10, 15, 20, 25, 30, 35, and 40 minutes during each 40-minute intervention session.
  The investigators will compare changes in systolic and diastolic blood pressure between the curated music playlist and guided mindfulness interventions using an automated oscillometric upper arm blood pressure monitor with measurements taken in triplicate at 5-minute intervals.
Changes in Heart Rate | 0, 5, 10, 15, 20, 25, 30, 35, and 40 minutes during each 40-minute intervention session.
  The investigators will compare changes in heart rate between the curated music playlist and guided mindfulness interventions using an automated oscillometric upper arm blood pressure monitor with measurements taken in triplicate at 5-minute intervals.

SECONDARY OUTCOMES:
Changes in Beat-to-Beat Blood Pressure (Finapres NOVA) | 0 to 40 minutes during each 40-minute intervention session.
  Continuous beat-to-beat blood pressure will be recorded using Finapres NOVA monitoring technology (Finapres Medical Systems, Netherlands) to allow for more detailed characterization of the cardiovascular response to music and mindfulness, potentially capturing effects on systolic and diastolic blood pressure not detected by periodic arm-cuff measurements.
Changes in Heart Rate (Finapres NOVA, Electrocardiogram-derived) | 0 to 40 minutes during each 40-minute intervention session.
  Heart rate will be recorded continuously using the electrocardiogram (ECG) channel of the Finapres NOVA, a non-invasive continuous hemodynamic monitoring technology (Finapres Medical Systems, Netherlands). Heart rate values will be derived from the ECG signal. This will allow for more detailed characterization of the cardiovascular response to music and mindfulness, potentially capturing effects on heart rate not detected by periodic arm-cuff measurements.
Change from Baseline in STAI-Y 1 | Baseline and immediately after each of the two 40-minute intervention sessions during the single study visit.
  The investigators will measure changes in acute anxiety using the State-Trait Anxiety Scale (STAI) - State subscale (form Y1) before and after each intervention. The STAI consists of 20 participant-rated statements, from 1 to 4 (1= Not at all, 4= Very much so) regarding their current anxiety (state). A lower score corresponds to less severity of symptoms.
Barcelona Music Reward Questionnaire (BMRQ) | Baseline
  The Barcelona Music Reward Questionnaire (BMRQ) is a validated 20-item questionnaire used to assess individual differences in the rewarding aspects of music listening. Each item is a statement rated on a 5-point Likert scale (1 = "Completely Disagree" to 5 = "Completely Agree"). Higher scores indicate a greater sensitivity to music-related reward. The total and subscale scores will be used to determine whether the extent of music reward experienced by participants predicts the magnitude of cardiovascular impact.
MUSE questionnaire | Baseline
  The MUSE questionnaire includes two quantitative items assessing average weekly and daily hours of music listening, as well as three 5-point Likert scale items evaluating the subjective importance of music, frequency of listening, and preference for specific genres. It will be used to characterize participants' music listening habits and attitudes and their relationship to cardiovascular outcomes.
Mindfulness Adherence Questionnaire (MAQ) | Baseline
  The Mindfulness Adherence Questionnaire (MAQ) is designed to measure the quantity and quality of an individual's mindfulness practice. It includes two quantitative items assessing frequency of formal practice and average duration of each session, as well as ten 5-point Likert scale items evaluating quality of mindfulness practice and time spent being mindful in everyday life, outside of formal sessions. It will be used to evaluate participants' experience with mindfulness and its relationship to cardiovascular outcomes.
Modified Tellegen Absorption Scale (MODTAS) | Baseline
  The Modified Tellegen Absorption Scale (MODTAS) is a validated 34-item questionnaire designed to measure an individual's engagement or immersion in sensory or imaginative experiences. Each item is rated on a 5-point Likert scale. It will be used to explore whether individual differences in trait absorption predict responsiveness to music and mindfulness interventions.
Subjective Enjoyment (Visual Analogue Scale) | Immediately after each of the two 40-minute intervention sessions during the single study visit.
  The investigators will assess subjective enjoyment of each intervention using 10-point visual analogue scales (VAS) administered immediately following each session. Participants will rate their enjoyment on a horizontal scale ranging from 0 ("not at all enjoyable") to 10 ("extremely enjoyable"). Including these measures will allow for assessment of potential preference effects that could influence cardiovascular outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Greenway, MD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital, McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data and the small sample size, which poses a risk of participant identification, the data will not be shared.